CLINICAL TRIAL: NCT03503383
Title: Evaluation of Mental Health Status in Pregnant Women Complaining of Hypertension With Pregnancy
Brief Title: Evaluation of Psychological Status in Pregnant Women Complaining of Hypertension With Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mena Malak Saleeb Abdalla, Principal Investigator, Zagazig University
Other Study IDs: MAbdalla1
Record Dates: First submitted 2018-03-26; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Hypertension With Pregnancy
Keywords: Hypertension with pregnancy; anxiety; depression; preeclampsia; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Pre-Eclampsia; Psychological Well-Being | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled group: pregnant women without any medical disorders during pregnancy
  Interventions: Behavioral: Patient Health Questionnaire-9; Behavioral: Generalized Anxiety Disorder Scale (GAD-7)
- Diseased group: Patients complaining of hypertension with pregnancy
  Interventions: Behavioral: Patient Health Questionnaire-9; Behavioral: Generalized Anxiety Disorder Scale (GAD-7)

INTERVENTIONS:
Behavioral: Patient Health Questionnaire-9 — PHQ-9 for assessing and monitoring depression severity
  Other Names: PHQ-9 depression scale
Behavioral: Generalized Anxiety Disorder Scale (GAD-7) — to diagnose generalized anxiety disorder, the GAD-7 also proved to have good sensitivity and specificity as a screener for panic, social anxiety, and post-traumatic stress disorder
  Other Names: GAD-7

SUMMARY:
This study is a case controlled study comparing mental health status and some psychological impacts between two groups of patients first group is pregnant women without any other medical disorder during pregnancy,the second group is pregnant women complaining of hypertension with pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* Hypertensive pregnant women for diseased group
* Normal pregnancy with no medical disorders associated in controlled group
* singleton pregnancy
* spontaneous pregnancy
* patients who are not divorced or not widow

Exclusion Criteria:

* non-pregnant women
* any other associated medical disorder with pregnancy rather than Hypertension
* any known psychological or mental disorder prior to pregnancy
* non spontaneous pregnancy as those whom conceived by IVF
* Twin or more pregnancy
* patients who are divorced or widow

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study only includes pregnant women
Study Population: This study is comparing between two groups, first group is healthy pregnant women and second group is pregnant women with hypertension . Both groups are assessed for both Anxiety and Depresion disorders.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression Evaluation using Patient Health Questionnaire-9 (PHQ-9) | 6 months
  Patient Health Questionnaire-9 is used to assess number of participants with depression.
Anxiety Evaluation using Generalized Anxiety Disorder Scale-7 (GAD-7) | 6 months
  Generalized Anxiety Disorder Scale (GAD-7) is used to assess number of participants with anxiety disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Mena M Abdalla, MSc, Principal Investigator — Zagazig University
Locations (2):
- Egypt (2):
  - Minya Health Insurance Hospital, Minya
  - Zagazig University Hospitals, Zagazig

IPD SHARING:
Plan to Share IPD: Undecided